CLINICAL TRIAL: NCT04951882
Title: Transplatation of Human Umbilcal Cord Derived Mesenchyamal Stem Cells in Acute Lung Injury: a Single Center Prospective Clinical Research
Brief Title: Application of hUC-MSCs in Treating Acute Lung Injury: a Single Center Prospective Clinical Research
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-592
Record Dates: First submitted 2021-06-08; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hUC-MSCs treatment (Placebo Comparator): Patients of acute lung injury will be treated by suspention of hUC-MSCs and albumin combined with standard therapies.
  Interventions: Biological: human derived umbilical cord derived mesenchymal stem cells
- non-cell therapy (No Intervention): Patients of acute lung injury will be treated by vehicle (albumin) combined with standard therapies.

INTERVENTIONS:
Biological: human derived umbilical cord derived mesenchymal stem cells — intravenous transplantation of human derived umbilical cord derived mesenchymal stem cells
  Arms: hUC-MSCs treatment

SUMMARY:
The patients suffered from acute lung ininjury (200<PaO2/FiO2 ≤ 300) will be divided into two groups: MSCs-treated group: patients are treated by intravenous injection of hUC-MSCs suspention ; control group: patients were treated with vehicle(Albumin) . The standard Therapies of acute lung injury were the same in both groups. In the following-up days, all the patients were monitored by the same items to evaluate the therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* 1.≤ 3 days (72h)
* 2.Age ≥18 years, ≤65 years
* 3.200<PaO2/FiO2 ≤ 300
* 4.Chest X-ray/chest CT : infiltrates of both lungs
* 5.Need assisted ventilation (ventilation or high flow oxygen therapy)
* 6.No left heart failure, pulmonary edema
* 7.Agree to participate and signe an informed consent

Exclusion Criteria:

* 1.Life expectancy <3 months due to non-respiratory failure
* 2.Patients receiving extracorporeal membrane oxygenation support therapy(ECMO),high frequency oscillatory ventilation
* 3.History of HIV, malignant tumors, or impaired immune function
* 4.Patients accepted major surgery in the past 14 days (such as tumor removal, thoracotomy, heart surgery, abdominal surgery, intracranial surgery, or surgery for more than 3 hours, etc.)
* 5.Pregnancy
* 6.Have a serious concomitant disease
* 7.Unable to follow-up
* 8.History of severe allergic reactions or allergy to saline and serum
* 9.Already participated in another clinical study within 12 weeks
* 10.Pulmonary edema caused by other underlying diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 | Day 3
  Oxygenation index
PaO2/FiO2 | Day 7
  Oxygenation index
PaO2/FiO2 | Day 14
  Oxygenation index
PaO2/FiO2 | Day 28
  Oxygenation index

SECONDARY OUTCOMES:
the days of ventialtion and hospital stay | Day 3
  the length of ventilation and hospital stay
the days of ventialtion and hospital stay | Day 7
  the length of ventilation and hospital stay
the days of ventialtion and hospital stay | Day 14
  the length of ventilation and hospital stay
the days of ventialtion and hospital stay | Day 28
  the length of ventilation and hospital stay

OTHER OUTCOMES:
IL-6 | Day 1
  inflammatory factors
IL-6 | Day 7
  inflammatory factors
IL-6 | Day 14
  inflammatory factors
IL-6 | Day 28
  inflammatory factors
IL-8 | Day 1
  inflammatory factors
IL-8 | Day 7
  inflammatory factors
IL-8 | Day 14
  inflammatory factors
IL-8 | Day 28
  inflammatory factors
TNF-a | Day 3
  inflammatory factors
TNF-a | Day 7
  inflammatory factors
TNF-a | Day 14
  inflammatory factors
TNF-a | Day 28
  inflammatory factors

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZU, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No